CLINICAL TRIAL: NCT00950066
Title: Study to Evaluate the Safety and Efficacy of Two Fixed Dose Combinations of Irbesartan / Amlodipine and Monotherapy After Eight Weeks of Treatment in Subjects With Uncomplicated Mild to Moderate Essential Hypertension
Brief Title: Irbesartan and Amlodipine Combination in Controlling Blood Pressure
Acronym: I-COMBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRBES_R_04320
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- Placebo (Placebo Comparator): Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with placebo once a day.
  Interventions: Drug: Placebo
- Irbesartan 150mg (Active Comparator): Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with Irbesartan 150 mg once a day.
  Interventions: Drug: IRBESARTAN (SR47436)
- Irbesartan 150 mg / Amlodipine 5 mg (Active Comparator): Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with Irbesartan 150 mg / Amlodipine 5 mg once a day.
  Interventions: Drug: Irbesartan / Amlodipine
- Amlodipine (Active Comparator): Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with Amlodipine 5 mg once a day.
  Interventions: Drug: Amlodipine
- Irbesartan 300 mg (Active Comparator): Active Comparator: Irbesartan
  Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with Irbesartan 300 mg once a day.
  Interventions: Drug: IRBESARTAN (SR47436)
- Irbesartan 300 mg / Amlodipine 5 mg (Active Comparator): Before randomization (common with other arms):
  There is an initial washout (placebo run-in) period of 2 weeks for subjects already on anti-hypertensive monotherapy.
  After randomization:
  8 weeks of treatment with Irbesartan 300 mg / Amlodipine 5 mg once a day.
  Interventions: Drug: Irbesartan / Amlodipine

INTERVENTIONS:
Drug: IRBESARTAN (SR47436) — Oral administration of Irbesartan 150mg or 300mg once a day
  Arms: Irbesartan 150mg; Irbesartan 300 mg
Drug: Amlodipine — Oral administration of Amlodipine 5mg once a day
  Arms: Amlodipine
Drug: Irbesartan / Amlodipine — Oral administration of Irbesartan 150 mg / Amlodipine 5mg or Irbesartan 300mg / Amlodipine 5mg once a day
  Arms: Irbesartan 150 mg / Amlodipine 5 mg; Irbesartan 300 mg / Amlodipine 5 mg
Drug: Placebo — Oral administration of a placebo once a day
  Arms: Placebo

SUMMARY:
The primary objective is to compare the extent of reduction of mean Seated Diastolic Blood Pressure (SeDBP) at the end of 8 weeks between each Fixed Dose Combination (FDC), its individual constituents administered as monotherapy and placebo.

The secondary objectives are:

* to compare the reduction of mean Seated Systolic Blood Pressure (SeSBP) at the end of 8 weeks from baseline between each FDC, its individual constituents administered as monotherapy and placebo.
* to compare the reduction of mean SeDBP and SeSBP at 4 weeks from baseline between each FDC, its individual constituents administered as monotherapy and placebo.

ELIGIBILITY:
Inclusion criteria:

* Subjects with uncomplicated mild to moderate essential hypertension (as per European Society of Cardiology Classification of Hypertension)

  * Treatment naïve subjects (newly diagnosed subjects or subjects currently only on lifestyle modification) with mean SeDBP of 95 to 109 mmHg at both screening and randomization visit (mean of 3 recordings at intervals of 1 minute) Or
  * Uncontrolled on any anti-hypertensive monotherapy and with mean SeDBP of 90 to 109 mmHg at screening and mean SeDBP of 95 to 109 mmHg at the randomization visit (mean of 3 recordings at intervals of 1 minute).
* Signed written informed consent obtained prior to inclusion in the study.
* Subjects willing to adhere to protocol and study requirements during the entire study duration.
* Subjects having no abnormalities in general physical examination.

Exclusion criteria:

* Subjects who are incapable of giving informed consent for the study.
* Subjects with SeDBP > or = 110mmHg and / or SeSBP > or = 180 mmHg measured at Doctor's office during screening or randomization visit
* Subjects having a difference of > 8 mmHg between any 2 of the 3 SeDBP measurements either at screening or at randomization.
* Subjects who are on any anti-hypertensive therapy and unable to discontinue the anti-hypertensive therapy safely for a period of at least 2 weeks as required by the protocol.
* Subjects who cannot be discontinued on medications prohibited by the protocol.
* Subjects on combination therapies for treatment of hypertension.
* Subjects with known documented secondary hypertension including (but not limited to) hypertension secondary to coarctation of aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.
* Subjects with known diabetes (Type 1 or Type 2).
* Subjects with known documented complications of hypertension including (but not limited to):

  * Cardiovascular disease: Ischemic heart disease (angina, myocardial infarction), heart failure, peripheral vascular disease.
  * Cerebrovascular disease: Stroke, cerebral hemorrhage.
  * Ophthalmic: Retinal hemorrhage, impaired vision, retinal microaneurysms.
* Subjects with known severe renal impairment (creatinine clearance < 30 ml/min) calculated using the Cockcroft-Gault equation.
* Subjects with hyperkalemia (>5.1mmol/L) and/or hyponatremia (<133mmol/L).
* Subjects with known severe hepatic impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal or history of hepatic encephalopathy, esophageal varices, or portocaval shunt.
* Subjects with clinically significant abnormalities on ECG
* Subjects with any other clinical condition which, in the opinion of the Investigator, might interfere with administration of Irbesartan or Amlodipine and evaluation of the study objectives.
* Subjects with known history of allergy considered due to any of the study drugs or their components, including excipients (lactose) and preservatives.
* Subjects with known history of substance abuse (drug or alcohol dependency, alcohol, if not stopped, <20gms per day will be allowed during the study period).
* Subjects known positive for HIV 1 or 2 virus.
* Subjects with known or suspected impairment of the immune function, and/or receiving immunosuppressive therapy, or having received immunosuppressive therapy within 30 days prior to study entry.
* Subjects who have received any other investigational drug within 30 days before inclusion.
* Pregnant (demonstrating a positive serum (ß-HCG) pregnancy test at screening visit) or lactating female subjects.
* Subjects and partners unwilling to employ adequate contraception during the course of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean change in SeDBP between each FDC, its individual constituents administered as monotherapy and placebo | At week 0, week 2, week 4 and week 8

SECONDARY OUTCOMES:
Difference in mean change in SeSBP between each FDC, its individual constituents administered as monotherapy and placebo | At week 0, week 2, week 4 and week 8
Difference in mean change in SeDBP and SeSBP between each FDC, its individual constituents administered as monotherapy and placebo | At week 0, week 2, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Aggarwal, MD, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan